CLINICAL TRIAL: NCT01980706
Title: Efficacy and Safety of High Dose Baclofen for Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-1743; 4R01AA020824-04 (NIH)
Record Dates: First submitted 2013-10-28; First posted 2013-11-11 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2018-10

CONDITIONS: Alcoholism
Keywords: Baclofen; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Baclofen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will take placebo for 16 weeks, 3 times per day. Placebo will be given in blister packs.
  Interventions: Drug: Placebo
- 30 Mg Baclofen (Active Comparator): Participants will take baclofen/placebo for 16 weeks, 3 times per day. Baclofen will be given in blister packs. The 30 mg/d arm will reach 30 mg/d at day 3 and titrate down starting at day 101.
  Interventions: Drug: Baclofen
- 90 mg Baclofen (Active Comparator): Participants will take baclofen/placebo for 16 weeks, 3 times per day. Baclofen will be given in blister packs. The 90 mg/d arm will reach 90 mg/d at day 12 and titrate down starting at day 95.
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen — Baclofen is a GABA-B agonist
  Other Names: Lioresal
  Arms: 30 Mg Baclofen; 90 mg Baclofen
Drug: Placebo — Pill containing no pharmacologically active substance.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The proposed study will carefully test the hypothesis that a robust dose of baclofen (90 mg/day) has efficacy and is safe in individuals with alcohol dependence. Furthermore, the proposal will test whether an indicator of physical dependence, i.e. drinks/drinking day, predicts response to baclofen. Additionally, the proposal will examine the anti-anxiety effects of baclofen within an alcohol dependent population and ascertain whether baseline levels of anxiety predict response to baclofen.

DETAILED DESCRIPTION:
Alcohol dependence (AD) is a common problem with significant health consequences. Treatment of AD is evolving to include both counseling methods and medications. Several medications have been discovered, that show efficacy in AD, e.g. naltrexone, acamprosate. However, the overall effect of existing medications is modest leaving a clear need for the development of new pharmacotherapies. The gamma-aminobutyric acid (GABA)-B receptor agonist baclofen has attracted attention as a potential new medication for AD based on preclinical data and early clinical trials. Baclofen is an FDA approved medication with an excellent safety profile even for patients with liver cirrhosis-a not uncommon consequence of AD. Questions have arisen with regards to the efficacy of baclofen and whether higher doses of baclofen are safe and more effective than the prior tested dose of 30 mg/ day. There is emerging evidence that severity of dependence is positively associated with baclofen response. The main goal of the present proposal is to test the efficacy and safety of 30 mg/d and 90 mg/d of baclofen compared to placebo controlling for severity of dependence as assessed by drinks/drinking day. A primary secondary goal will examine for an anxiolytic effect of baclofen. The study proposes to enroll 120 men and women with AD in a randomized, placebo-controlled trial to include at least 60 individuals with more severe AD (≥14 drinks/drinking day for men; ≥10 drinks/drinking day for women) with randomization to baclofen or placebo balanced for this variable. Baclofen will be titrated to 10 mg t.i.d over 3 days and to 30 mg t.i.d over 12 days and maintained at that level for 12 weeks and then downtitrated for a total study time of 16 weeks. Medical Management will be provided to encourage progress towards drinking goals and to enhance retention and compliance. Drinking patterns, anxiety levels, sleep patterns, craving for alcohol, gamma-glutamyl transferase (GGT) and carbohydrate deficient transferring (CDT) will be assessed. Trough blood levels of R & S-baclofen will be assessed in all individuals at week 4.

In summary, the present proposal is innovative and of clinical significance as it will test and compare standard and high-dose baclofen for efficacy and safety in individuals with AD. The proposal is adequately powered to test the primary hypothesis and provides good power to assess whether drinks/drinking day is predictive of baclofen response. Adequate power is also present to examine the anxiolytic effect of baclofen. Ascertaining the effects of standard and high-dose baclofen, the predictive value of heavy drinking on baclofen response and the anxiolytic effect of baclofen are important goals towards determining whether baclofen has true value for the clinical management of the patient with alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 65 meeting Diagnostic and Statistical Manual (DSM)-IV criteria for current alcohol dependence.
2. More than 14 drinks (women) or 21 drinks (men) per week including at least 2 heavy drinking days (men > 5 drinks/day; women > 4 drinks/day) per week in the 30-day period prior to screening. In addition we will recruit 50% of individuals who have a mean of ≥14 drinks/drinking day (men) or ≥10 drinks/drinking day (women) in the 30 days prior to screening.
3. Ability to understand and sign written informed consent.
4. Must have a 0.0 gms/dL breathalyzer reading on the day of screening and 0.0 gms/dL on the day of randomization.
5. Express a desire to achieve abstinence or to greatly reduce alcohol consumption
6. Must have a stable residence and be able to identify an individual who could contact participant if needed.

Exclusion Criteria:

1. Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern (e.g., renal insufficiency, cirrhosis, unstable hypertension, diabetes mellitus, seizure disorder). Clinically significant psychiatric illness including any psychotic disorder, bipolar disorder, severe depression, or suicidal ideation.
2. Other substance abuse or dependence disorder other than nicotine or alcohol or cannabis abuse.

   Occasional use of cocaine is acceptable.
3. Concurrent use of any psychotropic medication including antidepressants, mood stabilizers, antipsychotics, anxiolytics, stimulants, or hypnotics with the exception of stable doses of antidepressants for one month. Concurrent use of anticonvulsants, insulin, or oral hypoglycemics.
4. Prior history of adverse reaction to baclofen.
5. Creatinine level > Upper Limit of Normal (ULN) or Estimated Glomerular Filtration Rate < age norm.
6. aspartate aminotransferase (AST), or alanine transaminase (ALT) > 5 times ULN or bilirubin > 1.5 X ULN.
7. Positive urine toxicology screen with the exception of cannabis. Individuals with positive cannabis screens will be excluded only if they have a history of cannabis dependence.
8. Pregnant women and women of childbearing potential who do not practice a medically acceptable form of birth control (oral or depot contraceptive, or barrier methods such as diaphragm or condom with spermicidal).
9. Women who are breastfeeding.
10. Individuals requiring inpatient treatment or more intense outpatient treatment for their alcohol dependence.
11. Participation in any clinical trial within the past 60 days.
12. Court-mandated participation in alcohol treatment or pending incarceration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Garbutt, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 30 Mg Baclofen: Participants will take baclofen/placebo for 16 weeks, 3 times per day. Baclofen will be given in blister packs. The 30 mg/d arm will reach 30 mg/d at day 3 and titrate down starting at day 101.
  Baclofen: Baclofen is a gamma-aminobutyric acid (GABA)-B receptor agonist
Period: Overall Study
Arm/Group | Placebo | 30 Mg Baclofen | 90 mg Baclofen
Started | 40 | 43 | 37
Completed | 23 | 26 | 24
Not Completed | 17 | 17 | 13
Not completed — Withdrawal by Subject | 9 | 6 | 2
Not completed — Adverse Event | 1 | 2 | 5
Not completed — Lost to Follow-up | 3 | 4 | 3
Not completed — miscellaneous | 4 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 30 Mg Baclofen | 90 mg Baclofen | Total
Number analyzed (Participants) | 40 | 43 | 37 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (9.6) | 46.1 (10.4) | 44.8 (10.3) | 46.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 17 | 58
  Male | 20 | 22 | 20 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 6 | 14
  White | 36 | 36 | 30 | 102
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 43 | 37 | 120
Baseline Percentage of Heavy Drinking Days [Mean (Standard Deviation); unit: percentage of heavy drinking days] — Percentage of heavy drinking days over the prior 90 days
  percentage of heavy drinking days | 79 (21) | 73 (23) | 70 (26) | 74 (23)
Baseline Percentage of Abstinent Days [Mean (Standard Deviation); unit: Percentage of Abstinent Days] — Percentage of abstinent days over the prior 90 days.
  Percentage of Abstinent Days | 13 (17) | 17 (19) | 18 (20) | 16 (19)
Baseline Drinks/drinking day [Mean (Standard Deviation); unit: drinks per drinking day] | 9.3 (3.9) | 10.7 (7.7) | 10.0 (4.2) | 10.0 (5.6)
Goal of Abstinence [Count of Participants; unit: Participants] | 16 | 24 | 12 | 52
Craving for Alcohol [Mean (Standard Deviation); unit: units on a scale] — Penn Alcohol Craving Scale (PACS) is a five-item self administered instrument for assessing craving, frequency, intensity, and duration of thoughts about drinking as well as the ability to resist drinking. Scores range from a minimum of zero to a maximum of 30. Lower scores are associated with lower level of craving for alcohol.
  units on a scale | 14.5 (6.8) | 15.5 (7.2) | 15.3 (6.1) | 15.1 (6.7)
Carbohydrate Deficient Transferrin (CDT) [Mean (Standard Deviation); unit: % CDT] — laboratory measure that assesses levels of heavy drinking over time with greater specificity than gamma-glutamyl transferase (GGT). Population: Not all subjects had CDT analyzed.
  % CDT
    number analyzed (Participants) | 38 | 40 | 35 | 113
    (all) | 2.31 (1.95) | 1.72 (0.63) | 2.22 (1.46) | 2.07 (1.46)
Speilberger State Anxiety [Mean (Standard Deviation); unit: units on a scale] — The Spielberger State and Trait Anxiety Inventory (STAI) is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of state anxiety, which evaluates how the subject feels currently (transient anxiety). The State scale consists of 20 questions, each question rated 1-4, and a higher score indicates greater anxiety. Total score ranges from 20 (no anxiety) to 80 (maximum anxiety).
  units on a scale | 35.0 (10.5) | 36.3 (12.4) | 35.7 (9.7) | 35.7 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Heavy Drinking Days
Description: The frequency of heavy drinking days (5 or more drinks for a man and 4 or more drinks for a woman) as percentage during the treatment phase.
Time Frame: Every 1-2 weeks up to 16 weeks of active trial
Population: Post-randomization data were unavailable for 2 participants.
Measure: Least Squares Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | Placebo | 30 Mg Baclofen | 90 mg Baclofen
Number analyzed (Participants) | 40 | 42 | 36
percentage of heavy drinking days | 39 (4) | 42 (4) | 28 (4)
Statistical Analysis 1: Comparison: Placebo vs 30 Mg Baclofen vs 90 mg Baclofen; Test type: Superiority; p = 0.018, Mixed Models Analysis — Threshold for significance is <.05; Mean Difference (Net) = 4.16 — Overall, treatment effect F value testing under the null hypothesis the equality of the average outcome over the three groups

2. Primary Outcome: Mean Percentage of Abstinent Drinking Days
Description: Percent of abstinent days over the course of the trial.
Time Frame: Every 1-2 weeks up to 16 weeks of active trial
Population: Post-randomization data were unavailable for 2 participants.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | 30 Mg Baclofen | 90 mg Baclofen
Number analyzed (Participants) | 40 | 42 | 36
percentage of days | 47 (4) | 48 (4) | 59 (4)
Statistical Analysis 1: Comparison: Placebo vs 30 Mg Baclofen vs 90 mg Baclofen; Test type: Superiority; p = 0.028, Mixed Models Analysis — Threshold for significance is <.05; Mean Difference (Net) = 3.68 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Spielberger State-Trait Anxiety Inventory Score [State]
Description: The Spielberger State and Trait Anxiety Inventory (STAI) is a validated self-reporting instrument used to assess anxiety in adults.The inventory consists of state anxiety, which evaluates how the subject feels currently (transient anxiety). The State scale consists of 20 questions, each question rated 1-4, and a higher score indicates greater anxiety. Total score ranges from 20 (no anxiety) to 80 (maximum anxiety). The scores are averaged over the trial.
Time Frame: Every 1-2 weeks up to 16 weeks of active trial
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 30 Mg Baclofen | 90 mg Baclofen
Number analyzed (Participants) | 40 | 43 | 37
units on a scale | 35.2 (1.16) | 33.8 (1.12) | 33.6 (1.18)
Statistical Analysis 1: Comparison: Placebo vs 30 Mg Baclofen vs 90 mg Baclofen; Test type: Superiority; p = 0.52, Mixed Models Analysis — Threshold for significance is <.05; Mean Difference (Net) = 0.65 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Penn Alcohol Craving Scale Score
Description: Penn Alcohol Craving Scale (PACS) is a five-item self administered instrument for assessing craving, frequency, intensity, and duration of thoughts about drinking as well as the ability to resist drinking. Scores range from a minimum of zero to a maximum of 30. Lower scores are associated with lower level of craving for alcohol. Scores are averaged over the trial.
Time Frame: Every 1-2 weeks up to 16 weeks of active trial
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 30 Mg Baclofen | 90 mg Baclofen
Number analyzed (Participants) | 40 | 43 | 37
units on a scale | 10.1 (0.91) | 10.8 (0.88) | 9.4 (0.92)
Statistical Analysis 1: Comparison: Placebo vs 30 Mg Baclofen vs 90 mg Baclofen; Test type: Superiority; p = 0.43, Mixed Models Analysis — Threshold for significance is <.05; Mean Difference (Net) = 0.84 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Carbohydrate-deficient Transferrin
Description: Lab test assessing history of heavy drinking with greater specificity than GGT. Higher levels are indicative of greater levels of drinking.
Time Frame: End of trial, generally 16 weeks
Population: Post-randomization CDT was not collected for all participants.
Measure: Least Squares Mean (Standard Error); unit: % CDT
Arm/Group | Placebo | 30 Mg Baclofen | 90 mg Baclofen
Number analyzed (Participants) | 18 | 20 | 17
% CDT | 1.81 (.26) | 2.19 (.26) | 1.96 (.28)
Statistical Analysis 1: Comparison: Placebo vs 30 Mg Baclofen vs 90 mg Baclofen; Test type: Superiority; p = 0.60, ANCOVA — Threshold for significance is <.05; Adjusted for baseline; Mean Difference (Final Values) = 0.52 — Estimated parameter is the overall treatment main effect F statistic from the fitted ANCOVA model assessing the null hypothesis of equal values across the three groups

6. Other Pre Specified Outcome: Self-reported Sedation on at Least One Occasion by a Participant
Description: Any reporting of feeling sedated/sleepy/drowsy
Time Frame: Every 1-2 weeks up to 16 weeks of active trial
Population: Post-randomization data were unavailable for 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 30 Mg Baclofen | 90 mg Baclofen
Number analyzed (Participants) | 40 | 42 | 36
Participants | 14 | 25 | 20
Statistical Analysis 1: Comparison: Placebo vs 30 Mg Baclofen vs 90 mg Baclofen; Test type: Superiority; p = 0.07, Fisher Exact — Threshold for significance is <.05; Table probability for Fisher's Exact = .002

ADVERSE EVENTS:
Time Frame: Throughout treatment and for 4 weeks after treatment ended.
Arm/Group | Placebo | 30 Mg Baclofen | 90 mg Baclofen
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43 | 1/37
Other Adverse Events (participants affected / at risk) | 16/40 | 28/43 | 21/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | 30 Mg Baclofen (N=43) | 90 mg Baclofen (N=37)
Drowsiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Subject became very drowsy and fell asleep while driving though recovered and did not have an accident.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | 30 Mg Baclofen (N=43) | 90 mg Baclofen (N=37)
Sedation (Nervous system disorders) | 14 | 25 | 20 — Sleepiness, somnolence
Dizziness (Nervous system disorders) | 5 | 12 | 8 — Feeling dizzy
Itchiness/rash (Skin and subcutaneous tissue disorders) | 4 | 8 | 0
Fatigue/low energy (General disorders) | 2 | 5 | 2
Nausea (Gastrointestinal disorders) | 4 | 5 | 4
Constipation (Gastrointestinal disorders) | 3 | 4 | 2
Headache (General disorders) | 3 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT01980706/Prot_SAP_000.pdf